CLINICAL TRIAL: NCT00006490
Title: HIV-1 Resistance Testing During Antiretroviral Failure: Comparison of Sequencing Versus Phenotyping
Brief Title: A Comparison of Two Tests for Anti-HIV Drug Resistance
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5076; AACTG A5076
Record Dates: First submitted 2000-11-08; First posted 2001-08-31 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2004-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Resistance, Microbial; Sequence Analysis, DNA; Microbial Sensitivity Tests; Genotype; Phenotype; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to compare 2 different types of tests of the HIV virus to see which specific anti-HIV drugs would work the best.

Drug resistance is a major reason for therapy failure in HIV patients. Two types of tests can detect resistance to drugs: 1) genotyping (sequencing), which looks at the DNA sequence of a virus to see whether it has developed any genetic resistance; 2) phenotyping, which looks at the ability of different drugs to suppress virus growth in the laboratory. Genotyping and phenotyping can help doctors give patients the most effective drug therapy.

DETAILED DESCRIPTION:
The emergence of drug resistance is a major factor contributing to the failure of antiretroviral therapy in HIV-infected patients. Drug resistance can be detected by genotypic or phenotypic assays, both having distinct advantages and disadvantages. Results from genotypic and phenotypic testing are helpful in excluding from the subsequent regimen drugs to which the resistance is identified, and both tests predict virologic response to salvage therapy in patients who have failed a previous regimen. Resistance testing is likely to be beneficial as an aid in selecting a salvage regimen.

At entry, patients are randomized to Arm A (sequencing) or Arm B (phenotyping) and have a resistance test drawn while still receiving the current regimen even though regimen failure is suspected. The test results are available between Weeks 1 and 4, inclusive. There are weekly visits for the first 4 weeks after entry to monitor viral load and maintenance of the current failing (prestudy) regimen. If virologic failure is confirmed, a new regimen is chosen and prescribed at the first visit after resistance test results are available. [AS PER AMENDMENT 12/6/00: If the resistance assay fails to yield results, another regimen is chosen and prescribed based on the patient's medical and medication history.] If virologic failure is not confirmed, the current drug regimen is not changed. Otherwise, on-site study visits occur every 4 weeks until Week 24 and then every 8 weeks thereafter through Week 48. [AS PER AMENDMENT 12/6/00: on-site study visits occur every 4 weeks until Week 24 and then every 8 weeks thereafter]. Medical resource use is assessed at baseline and then every 8 weeks through Week 48. Quality of life is assessed at baseline and then every 16 weeks through Week 48.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have failed 2 to 4 anti-HIV regimens containing 3 or more combinations of drugs. A patient has failed his/her current regimen if he/she has, within 30 days of study entry, either a viral load (level of HIV in the blood) of at least 10,000 copies/ml or 2 tests which show a viral load between 1,000 and 10,000 copies/ml.
* Have taken 3 or more anti-HIV drugs for 8 or more weeks before the study.
* Are at least 14 years old.
* Have consent of parent or guardian if less than 18 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have failed only 1 anti-HIV drug combination.
* Have failed 5 or more anti-HIV drug combinations, each containing 3 to 5 drugs.
* Have had and received the results of prior resistance tests.
* Have had treatment with a combination of 6 or more anti-HIV drugs.
* Have problems absorbing food in the intestine.
* Have had HIV vaccines.
* Have taken drugs that affect the immune system or investigational drugs.
* Are taking medications not allowed with protease inhibitors (PIs) if PIs would be part of their anti-HIV treatment during the study.
* Have failed anti-HIV therapy due to nonadherence to medication.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600

CONTACTS AND LOCATIONS:
Overall Officials: Richard D'Aquila, Study Chair; Daniel Kuritzkes, Study Chair
Locations (47):
- United States (46):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - University of California San Francisco, San Francisco, California
  - Univ of California San Francisco, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown Univ / Miriam Hosp, Providence, Rhode Island
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - Julio Arroyo, West Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico